CLINICAL TRIAL: NCT00120588
Title: Effect of Magnesium Sulfate on the Incidence of Periventricular Leukomalacia in the Very Preterm Neonate
Brief Title: Neuroprotection by Magnesium Sulfate Given to Women at Risk of Very Preterm Birth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1997/575/HP
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Preterm Birth; Periventricular Leukomalacia; Brain Ischemia; Intracranial Hemorrhages
Keywords: brain protection; white matter injury; neurodevelopmental sequelae; magnesium sulfate; intraventricular hemorrhage
MeSH Terms: conditions — Premature Birth; Leukomalacia, Periventricular; Brain Ischemia; Intracranial Hemorrhages | interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: magnesium

SUMMARY:
Magnesium is neuroprotective in neonatal animal models of acquired hypoxic-ischemic and/or inflammatory cerebral lesions. It is associated with a significant reduction of perinatal death and cerebral palsy in some observational studies.

The objective of the study is to assess if prenatal magnesium sulfate given to women at risk of preterm birth before 33 week's gestation is neuroprotective.

DETAILED DESCRIPTION:
This is a randomized controlled trial at 18 french tertiary hospitals with stratification by center and multiple births in women at risk of preterm birth before 33 week's gestation and without vascular disease of pregnancy.

Women received 4 g of a 0.1 g/ml magnesium sulfate solution or isotonic serum chloride solution (0.9%).

The main outcome measures are rates of mortality up to discharge, of severe white matter injury (defined by the presence of cavitations and/or intraparenchymal haemorrhages on cranial ultrasonographic studies) and of combined death and severe white matter injury.

The secondary outcome measures are rates of white matter injury (defined by the presence of cavitations and/or intraparenchymal haemorrhages and persisting hypechogenicities at 15 day intervals on cranial ultrasonographic studies), follow-up at two years of age

ELIGIBILITY:
Inclusion Criteria:

* women pregnant with single, twin or triplet very preterm fetuses younger than 33 week's gestational age if birth was expected or planned within 24 hours

Exclusion Criteria:

* women with vascular disease of pregnancy
* women with severe malformation or chromosomal abnormalities in the fetus
* women with hypotension
* renal insufficiency
* cardiac rhythmic abnormalities
* intake of calcium channel inhibitors
* digitalis or indomethacin less than 24 hours
* persistence of signs of cardiovascular toxicity or tachycardia for more than one hour after cessation of betamimetic intake
* myasthenia
* emergency C section

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 1997-07; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
death up to discharge of hospital
severe white matter injury
combined death up to discharge and severe white matter injury

SECONDARY OUTCOMES:
white matter injury
cystic periventricular leukomalacia
topography of cysts
intraventricular/intraparenchymal haemorrhages
side effects of magnesium sulfate in mothers and preterm newborns
follow-up at two years of age

CONTACTS AND LOCATIONS:
Overall Officials: Stephane MARRET, MD-PhD, Principal Investigator — university; Stephane Marret, MD-PhD, Principal Investigator — University Hospital, Rouen; Jacques Benichou, MD-PhD, Study Director — University hopsital of Rouen
Locations (1):
- Charles-Nicolle hospital, Rouen, Normandy, France

REFERENCES:
- [Derived] Chollat C, Enser M, Houivet E, Provost D, Benichou J, Marpeau L, Marret S. School-age outcomes following a randomized controlled trial of magnesium sulfate for neuroprotection of preterm infants. J Pediatr. 2014 Aug;165(2):398-400.e3. doi: 10.1016/j.jpeds.2014.04.007. Epub 2014 May 14. PMID 24837863